CLINICAL TRIAL: NCT05526027
Title: Real-world Efficacy and Safety of CFTR Modulator Therapy in Adult Patients With Cystic Fibrosis
Brief Title: Real-world Efficacy and Safety of Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) Modulator Therapy in Adult Patients With Cystic Fibrosis (CF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Stefanie Vincken, Medical doctor, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUN1432021000472
Record Dates: First submitted 2022-08-18; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ETI (Other): pwCF which are CFTR-modulator naive and pwCF previously treated with a CFTR-modulator (i.e. tezacaftor-ivacaftor or lumacaftor-ivacaftor) will undergo standard-of-care examinations as well as examinations in the context of this trial (i.e. CFQ-R, PHQ-9, GAD-7 and SNOT-22 questionnaires, fecal elastase measurement)
  Interventions: Diagnostic Test: CFQ-R questionnaire, SNOT-22 questionnaire, fecal elastase measurement

INTERVENTIONS:
Diagnostic Test: CFQ-R questionnaire, SNOT-22 questionnaire, fecal elastase measurement — cf supra

SUMMARY:
In this trial real-world data on the safety (side effects and medication interactions) and efficacy (evolution of lung function testing, chronic bacterial airway infection, quality of life and endo- and exocrine pancreatic function) will be collected in adult people with cystic fibrosis (pwCF) eligible for elexacaftor-tezacaftor-ivacaftor (ETI) up until 2 years after the start of this therapy.

DETAILED DESCRIPTION:
PwCF group A: CFTR-modulator-naive pwCF eligible for ETI (based on age and CFTR genotype)

PwCF group B: pwCF already on CFTR modulating therapy (i.e. ivacaftor-lumacaftor or ivacaftor-tezacaftor) and switching to ETI.

Patients in both groups will undergo these examinations:

* Physical examination (including weight)
* Anamnesis for current and recent medication use (including dosage of pancreatic enzymes) and for acute respiratory exacerbations
* Lung function testing including spiometry, multiple breath washout testing and fractional exhaled nitric oxide
* Blood sampling: liver function tests, creatine kinase, albumin, PT, red and white blood cell count, platelet count
* Sputum/cough swab sampling
* fecal elastase measurement
* Cystic fibrosis questionnaire-revised (CFQ-R) questionnaire
* Patient health questionnaire-9 (PHQ-9) questionnaire
* General anxiety disorder-7 (GAD-7) questionnaire
* Sino-nasal outcome test-22 (SNOT-22) questionnaire

These will be performed at baseline (prior to the start of ETI, on the same day of start of ETI), and every 3 months (+/- 7 days) thereafter. A blood sample will also be performed 14 (+/- 7 days) days after start of ETI (for safety). Fecal elastase measurement will only be performed at baseline if not available in the patient's medical record, and only 6 months after start of ETI.

ELIGIBILITY:
Inclusion Criteria:

* eligible for ETI (i.e. age above 18 years and CFTR genotype F508del/any) based on reimbursement criteria in Belgium

Exclusion Criteria:

* inability to perform lung function testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
percent predicted forced expiratory volume in 1 second (ppFEV1) | 2 years
Lung clearance index (LCI) | 2 years
Fractional excretion of nitric oxide (FeNO) | 2 years
CFQ-R questionnaire | 2 years
fecal elastase (microgram per gram of feces) | 2 years
  the concentration of elastase (a pancreatic enzyme) in feces before and 6 months after start of CFTR modulating treatment, as a surrogate measure for pancreatic function
the amount of participants experiencing a treatment-related adverse event | 2 years
annual acute exacerbation rate | 2 years
body mass index (BMI) | 2 years

SECONDARY OUTCOMES:
SNOT-22 questionnaire | 2 years
GAD-7 questionnaire | 2 years
PHQ-9 questionnaire | 2 years
aerobic culture on sputum or cough swab sample | 2 years
dosage of pancreatic enzyme replacement therapy | 2 years

IPD SHARING:
Plan to Share IPD: No